CLINICAL TRIAL: NCT04842019
Title: An Open-label, Multi-center, Single-cohort, Post-marketing Phase 4 Study to Evaluate the Efficacy, Pharmacodynamics, and Safety of the Anti-FGF23 Antibody, KRN23, in Adult Chinese Patients With X-linked Hypophosphatemic Rickets/Osteomalacia
Brief Title: Study to Assess the Safety, Pharmacokinetics and Efficacy of KRN23 in Adult Chinese Patients With XLH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRN23-CN005; CTR20210506 (Other: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2021-03-30; First posted 2021-04-12 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: X-linked Hypophosphatemia (XLH)
MeSH Terms: conditions — Familial Hypophosphatemic Rickets | interventions — burosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KRN23 (Experimental): KRN23 1 mg/kg administered subcutaneously (SC) every 4 weeks for 48 weeks. Before KRN23 treatment, all patients will receive oral phosphate and vitamin D analogs for 12 weeks of Run-in period.
  Interventions: Drug: KRN23

INTERVENTIONS:
Drug: KRN23 — KRN23 is a sterile clear colourless and preservative free solution supplied in single use 5 mL vials containing 1 mL of KRN23 at a concentration of 30mg/mL
  Other Names: Burosumab; Crysvita

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics and efficacy of KRN23 in adult Chinese patients with XLH

ELIGIBILITY:
Inclusion Criteria:

1. Male or female Chinese patients, aged 18 to 65 years (inclusive) at the time of signing the ICF
2. Diagnosis of XLH supported by classic clinical features of adult XLH (such as short stature or bowed legs) and at least either of the following at screening:

   * Confirmed PHEX mutation (prior to the study with historic record) in the patient or a directly related family member with appropriate X linked inheritance
   * Serum iFGF23 level ≥30 pg/mL by the Kainos assay at Screening
3. Biochemical findings consistent with XLH following overnight fasting (≥8 hours) at Screening:

   * Serum phosphorus <2.5 mg/dL (0.81 mmol/L). Serum phosphorus level may be re tested (once only) at least 7 days after discontinuation of therapy, if applicable.
   * TmP/GFR of <2.5 mg/dL
4. Presence of skeletal pain attributed to XLH/osteomalacia, as defined by a score of ≥4 on the BPI Worst Pain question at Screening (Skeletal pain that, in the opinion of the investigator or subinvestigator, is attributed solely to causes other than XLH/osteomalacia [e.g., back pain or joint pain in the presence of severe osteoarthritis by radiograph in that anatomical location] in the absence of any skeletal pain likely attributed to XLH/osteomalacia should not be considered for eligibility)
5. Patients who are taking chronic pain medications (including narcotic pain medications/opioids) must be on a stable regimen for at least 21 days before signing the ICF and be willing to maintain the medications at the same stable dose(s) and schedule throughout the study. The dose must not exceed 60 mg oral morphine equivalents/day
6. Able to receive conventional therapy (oral phosphate and pharmacologic vitamin D [or metabolites/analogs])
7. Written informed consent provided after the nature of the study has been explained and prior to any research related procedures
8. Willing to provide access to prior medical records for the collection of biochemical and radiographic data and disease history
9. Have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study (female patients of child-bearing potential only)
10. Be willing to use an effective method of contraception while participating in the study (sexually active patients of child bearing potential) and for 12 weeks after last dose of study drug. Women of non child bearing potential are defined as permanently sterile (i.e. due to hysterectomy or bilateral oophorectomy) or postmenopausal (defined as at least 12 months postcessation of menses without an alternative medical cause). Postmenopausal status of female patients will be confirmed with a Screening serum follicle stimulating hormone (FSH) level >40 mIU/mL
11. Be willing and able to complete all aspects of the study, adhere to the study visit schedule, and comply with the assessments, as judged by the investigator or subinvestigator
12. Have completed entries for ≥4 of 7 consecutive days of the patient diaries before Week -14

Exclusion Criteria:

1. Use of a pharmacologic vitamin D, its metabolites, or analogs, and oral phosphate for treatment of XLH within 14 days prior to Screening.
2. Use of aluminum hydroxide antacids, acetazolamide, thiazide diuretics and/or systemic corticosteroids within 14 days prior to Week -14
3. Corrected serum calcium level ≥10.8 mg/dL (2.69 mmol/L) at Screening
4. Plasma iPTH ≥2.5 times the upper limit of normal at Screening
5. Uncontrolled diabetes mellitus, defined as HbA1c >7.5% at Screening
6. Use of medication to suppress PTH (e.g., Sensipar®, cinacalcet, calcimimetics) within 60 days before signing the ICF
7. Use of oral bisphosphonates in the 2 years before signing the ICF
8. Planned or recommended orthopedic surgery within the clinical trial period
9. History of traumatic fracture or orthopedic surgery within 6 months before signing the ICF
10. Use of KRN23, or any other therapeutic mAb within 90 days before signing the ICF
11. Use of any investigational product or investigational medical device within 30 days before signing the ICF, or requirement for any investigational agent prior to completion of all scheduled study assessments
12. Pregnant or breastfeeding at Screening or Week -14, or intention to become pregnant (the patient or partner) at any time during the study
13. Unable or unwilling to withhold prohibited medications throughout the study
14. Presence or history of any hypersensitivity, or allergic or anaphylactic reactions to any mAb or KRN23 excipients that, in the judgment of the investigator or subinvestigator, places the patient at increased risk for adverse effects
15. Positive for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibody at Screening, or prior history of positive test
16. History of recurrent infection or predisposition to infection, or of known immunodeficiency
17. Presence of malignant neoplasm (except basal cell carcinoma)
18. Presence of a concurrent disease or condition that would interfere with study participation or affect safety
19. Presence or history of any condition that, in the view of the investigator or subinvestigator, places the patient at high risk of poor treatment compliance or of not completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-08-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (CFB) in mean serum phosphorus level at the end of the dose cycle | Weeks 4, 8, 12, 16, 20, 24, 36, and 48

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) Worst Pain score over time | Weeks 0, 12, 24, 36, and 48
  Change from baseline to post-baseline visits in BPI-Q3 (Worst Pain) score as averaged from daily diary scores recorded over 1 week and the study visit score. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Question 3 of the short-form BPI (BPI-Q3) asks subjects to rate their pain at its worst in the last 24 hours on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change in BPI Pain Severity score and Pain Interference score over time | Weeks 0, 12, 24, 36, and 48
  Change from baseline to post-baseline visits in BPI pain severity score as averaged from daily diary scores recorded over 1 week and the study visit score. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). The severity of pain in the last 24 hours is rated on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Change in BPI Pain Interference score over time | Weeks 0, 12, 24, 36, and 48
  Change from baseline to post-baseline visits in BPI pain interference score as recorded on the day of the study visit. The BPI evaluates the condition of all pain over the previous 24 hours. Two dimensions are measured: pain severity (worst, least, average, and now) and the impact of pain on functioning (pain interference with general activity, walking, work, mood, enjoyment of life, relations with others, and sleep). Pain interference in the last 24 hours is rated on a scale of 0 (does not interfere) to 10 (completely interferes).
Change in the Stiffness and Physical Function domains of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) over time | Weeks 0, 12, 24, 36, and 48
  The WOMAC is a 24-item participant-reported questionnaire with two domains, Stiffness (2 questions) and Physical Function (17 questions) over the previous 48 hours. The WOMAC is administered in a 5-point Likert-scale format using descriptors of none, mild, moderate, severe, and extreme corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse stiffness and functional limitations. Scores are normalized to a 0-100 metric where 0 was the best health state and 100 the worst.
Change in the health related QOL assessment by Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function over time | Weeks 0, 12, 24, 36, and 48
  The PROMIS was developed by the National Institutes of Health and uses domain-specific measures to assess patient well-being (Broderick et al. 2013), (NIH 2015). It uses a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For the Physical Function Domain, increases indicate greater mobility.
The proportion of subjects achieving mean serum phosphorus levels above the lower limit of normal (LLN; 2.5 mg/dL [0.81 mmol/L]) at the end of the dosing cycle | Weeks 4, 8, 12, 16, 20, 24, 36, and 48
The proportion of subjects achieving mean serum phosphorus levels above the LLN (2.5 mg/dL [0.81 mmol/L]) at the mid-point of dosing cycle | Weeks 2, 6, 10, 14, 18 and 22
CFB in mean serum phosphorus level at the mid-time point of dosing cycle | Weeks 2, 6, 10, 14, 18 and 22
Mean percent CFB in serum phosphorus levels averaged at the end of dose cycles | Baseline to Week 48
Cumulative exposure: area under curve (AUC) of serum phosphorus | Baseline to Week 48
Change in serum 1,25(OH)2D over time | Baseline to Week 48
Change in urinary phosphorus over time | Baseline to Week 48
Change in ratio of renal tubular maximum reabsorption rate of phosphate to glomerular filtration rate (TmP/GFR; algorithm method) over time | Baseline to Week 48

OTHER OUTCOMES:
Radiologic healing or resolution of pre-existing fractures and/or pseudofractures, as defined by skeletal survey at Baseline and subsequent targeted radiography | Weeks 0, 12, 24, 36, and 48
Change in enthesopathy spur at the calcaneus measured by lateral foot X-rays | Weeks 0, 24 and 48
Change in 6-minute walking test (6MWT) over time | Weeks 0, 12, 24, 36, and 48
Safety of KRN23 by studying the number, severity and relatedness of Adverse Events (including laboratory and imaging assessments) | Week 0 to Week 56
  Incidence, frequency, and severity of AEs and SAEs, including clinically significant changes in laboratory assessments as well as ECHO, ECG, ultrasound, vital sign, X-Ray images and Anti-KRN23 antibody.
Pharmacokinetics: KRN23 concentrations | Week 0, 1, 2, 4, 21, 22, 24, 36, 48 and 56
  KRN23 concentration in the Mid and end of dose cycles.
Change from Week -14 to Baseline in serum phosphorus over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in serum phosphorus over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in serum 1,25(OH)2D over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in serum 1,25(OH)2D over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in plamas iPTH over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in plamas iPTH over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in serum calcium over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in serum calcium over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in urinary phosphorus over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in urinary phosphorus over time during Run-in Period | Week -14, -10 and -4
Change from Week -14 to Baseline in TmP/GFR over time during Run-in Period | Week -14, -10 and -4
Percent change from Week -14 to Baseline in TmP/GFR over time during Run-in Period | Week -14, -10 and -4
Safety of conventional therapy by studying the number, severity and relatedness of Adverse Events | Week -14 to Week 0
  Incidence, frequency, and severity of AEs and SAEs, including clinically significant changes in laboratory assessments during Run-in period

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Peking Union Medical College Hospital, Beijing
  - The First Medical Center of Chinese People's Liberation Army General Hospital, Beijing
  - Nanfang Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Shanghai 6th Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No